CLINICAL TRIAL: NCT03670784
Title: Incidence and Trend of Ectopic Pregnancy 2009-2018 - A Population-based Study
Brief Title: Occurrence and Trend of Pregnancies Growing Outside the Womb (Ectopic Pregnancy) 2009-2018. A Study on a Defined Group of Persons
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20257
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Pregnancy, Ectopic
Keywords: Ectopic pregnancy; Electronic medical records; Chart Review; Intrauterine device (IUD)
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women_KPNC: Women of reproductive age who are enrolled in the US-health plan Kaiser Permanente Northern California (KPNC).
  Interventions: Other: No intervention
- Women_KPSC: Women of reproductive age who are enrolled in the US-health plan Kaiser Permanente Southern California (KPSC).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, epidemiological investigation

SUMMARY:
In this trial researchers want to learn more about the occurrence of pregnancies growing outside the womb over the last decade (2009-2018) and the potential risk factors associated with pregnancies growing outside the womb. Electronic data in women who were age 15 to 44 years abstracted from health care systems such as electronic health records (EHR), regional claims systems and administrative databases were used to address research questions on ...

* occurrence and trends of pregnancies growing outside the womb;
* influence of method of contraception used on occurrence and trends of pregnancies growing outside the womb;
* potential risk factors associated with pregnancies growing outside the womb;
* trends in management of pregnancies growing outside the womb over the last decade.

DETAILED DESCRIPTION:
The overall goal of this study is to assess the incidence rate of ectopic pregnancy over the last decade in a representative population of US women and potential risk factors associated with ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women of age 15 to 44 years between 01-Jan-2009 and 31-Dec-2018
* Women enrolled in health plans Kaiser Permanente Northern California (KPNC) and Kaiser Permanente Southern California (KPSC)
* Women with at least 12 months membership in KPNC and KPSC prior to enrollment

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Health-insured women of reproductive age from California (USA)
Sampling Method: Non-Probability Sample
Enrollment: 3922877 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Number of ectopic pregnancies | Retrospective analysis of data from 2009 to 2018
  Overall and during contraceptive use
Person-time at risk | Retrospective analysis of data from 2009 to 2018
  Person-time at risk is the time without ectopic pregnancy [in years, months, or days] that all subjects contributed to the study since enrollment.
Number of ectopic pregnancies | Retrospective analysis of data from 2009 to 2019
  During contraceptive and non- contraceptive use

SECONDARY OUTCOMES:
Risk factors for ectopic pregnancies | Retrospective analysis of data from 2009 to 2018
  Investigated risk factors comprise various demographic and clinical factors, contraceptive use and reproductive factors.
Accuracy of electronic health data to identify diagnosis of ectopic pregnancy | Retrospective analysis of data from 2009 to 2018
  Assessment by chart review of random samples of 0.001% of women per site and year.
Accuracy of electronic health data to identify contraceptive method at time of diagnosis of ectopic pregnancy | Retrospective analysis of data from 2009 to 2018
  Assessment by chart review of random samples of 0.001% of women per site and year.
Accuracy of electronic health data to identify contraceptive method over time | Retrospective analysis of data from 2009 to 2018
  Assessment by chart review of random samples of 0.001% of women per site and year.
Accuracy of electronic health data to identify induced abortions | Retrospective analysis of data from 2009 to 2018
  Assessment by chart review of random samples of 0.001% of women per site and year.
Numbers of ectopic pregnancies managed surgically | Retrospective analysis of data from 2009 to 2018
Numbers of ectopic pregnancies managed medically | Retrospective analysis of data from 2009 to 2018
Risk factors for ectopic pregnancies | Retrospective analysis of data from 2009 to 2019
  Risk factors will be investigated in women with current contraceptive use and non-contraceptive
Accuracy of the contraceptive algorithm | Retrospective analysis of data from 2009 to 2019
  Trained abstractors will conduct chart reviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com